CLINICAL TRIAL: NCT01085747
Title: Covered Self-expandable Metal Stents Versus Multiple Plastic Stents for Benign Biliary Stricture Caused by Chronic Pancreatitis: a Prospective Randomized Study
Brief Title: Endoscopic Treatment of Biliary Stricture Caused by Chronic Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Turku (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Halttunen Jorma, Jorma Halttunen, MD, PhD, Helsinki University Central Hospital
Other Study IDs: 98/13/03/03/08
Record Dates: First submitted 2010-03-08; First posted 2010-03-12 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Biliary Stricture; Chronic Pancreatitis
Keywords: Chronic pancreatitis; Biliary stricture; Endoscopic treatment; SEMS
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Plastic stent
- Covered SEMS

SUMMARY:
Benign biliary strictures can be endoscopically treated with plastic or self-expandable metal stents (SEMS). The purpose of the prospective randomized study is to compare the safety and feasibility of covered SEMS with multiple plastic stents in the treatment of benign biliary stricture caused by chronic pancreatitis.

DETAILED DESCRIPTION:
All consecutive patients admitted for ERCP and treated for benign biliary stricture caused by chronic pancreatitis are prospectively enrolled in the study.

At the initial ERCP, an endoscopic sphincterotomy will be performed and one 10 Fr plastic stent will be inserted for the initial treatment of cholestasis in all patients.Pancreatic stent will be inserted if indicated. One to three months after the initial ERCP the patients will be randomized into two groups: those who receive cSEMS and those who receive multiple plastic stents into the bile duct. For the randomization, sealed envelopes will be used. As for cSEMSs, removable cSEMSs with diameter of 10 mm will be placed. A dilation with a 8-10mm balloon will be performed before and after the stent placement to secure the stent expansion. As for plastic stents, minimum three simultaneous 10 Fr stents will be inserted after 8-10 mm balloon dilation.

After three months a further ERCP will be performed. The number of plastic stents will be increased maximally to six 10 Fr stents after dilation if possible. In the group with cSEMS, the position of the stent will be controlled.

Once the cSEMS or plastic stents have been in place for minimum six months, the stents will be removed at the last ERCP.

Follow-up

Clinical response (adequate biliary drainage) is the primary endpoint of the study. Therefore, blood liver function tests (bilirubin, alkaline phosphatase) as well as the minimum diameter of the common bile duct in the area of the stricture, the maximum diameter of the common bile duct above the stricture and the length of the stricture are measured at ERCPs at the time of the initial plastic stent insertion (i.e. the first ERCP) and at removal of cSEMS or multiple plastic stents (the last ERCP). In addition, blood liver function tests are measured and abdominal ultrasonography performed in the follow-up six months and two years after the stent removal.

Morbidity and mortality are additional endpoints of the study. Therefore, complications (deaths, stent occlusions, dislodgements or migrations, cholangitis, hemobilia, stone formation above the stent), management of complications, admission times, surgical interventions and any additional care needed are monitored and recorded during the follow-up time. Patients are asked to contact the physician at any time if symptoms such as fever, abdominal pain or jaundice occur.

ELIGIBILITY:
Inclusion Criteria:

* Benign biliary stricture caused by chronic pancreatitis

Exclusion Criteria:

* Malignancy, cirrhosis acute/chronic hepatitis or abnormal hepatic imaging. First attack of acute pancreatitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients admitted for ERCP and treated for benign biliary stricture caused by chronic pancreatitis are prospectively enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2013-05 (Actual); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Stricture resolution of the common bile duct in the two study groups | 2.5 years
  Stricture resolution during stenting and follow-up period, defined by normal liver function tests and abdominal ultrasonography

SECONDARY OUTCOMES:
Stent removability | Time from stent removal to 1 month post-stent removal
  Ability to remove stents endoscopically after six months without stent-removal related complications
Occurrence of complications related to stents and procedure | 2.5 years
Length of endoscopic procedures in the two groups | All endoscopic procedures

CONTACTS AND LOCATIONS:
Overall Officials: Jorma Halttunen, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Haapamaki C, Kylanpaa L, Udd M, Lindstrom O, Gronroos J, Saarela A, Mustonen H, Halttunen J. Randomized multicenter study of multiple plastic stents vs. covered self-expandable metallic stent in the treatment of biliary stricture in chronic pancreatitis. Endoscopy. 2015 Jul;47(7):605-10. doi: 10.1055/s-0034-1391331. Epub 2015 Jan 15. PMID 25590182